CLINICAL TRIAL: NCT02298192
Title: A Clinical Trial Comparing Efficacy and Safety of Insulin Degludec/Liraglutide (IDegLira) in Subjects With Type 2 Diabetes Mellitus Using Two Different Titration Algorithms
Acronym: DUAL™ VI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-4056; 2012-004625-25 (EudraCT Number); U1111-1135-6634 (Other: WHO)
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Once weekly titration (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- Twice weekly titration (Experimental)
  Interventions: Drug: insulin degludec/liraglutide

INTERVENTIONS:
Drug: insulin degludec/liraglutide — For subcutaneous (s.c., under the skin) injection, once daily. Subjects will be instructed to continue with the same dose of OADs (metformin alone or in combination with pioglitazone), as prior to the trial.

SUMMARY:
This trial is conducted in Europe, North America and the United States of America.

The aim of this trial is to compare two different titration algorithms of insulin degludec/liraglutide.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Male or female equal to or above 18 years of age
* HbA1c (glycosylated haemoglobin) 7.0 - 10.0% [53 mmol/mol - 86 mmol/mol] (both inclusive), confirmed by the central laboratory
* Stable daily treatment with metformin (above or equal to 1500 mg or max tolerated dose) with or without pioglitazone (above orequal to 30 mg) for at least 90 days prior to screening
* Body Mass Index (BMI) below or equal to 40 kg/m^2

Exclusion Criteria:

* Current use of any anti-diabetic drugs (except for metformin and pioglitazone) or anticipated change in concomitant medication, which, in the opinion of the investigator, could interfere with the glucose metabolism (e.g. systemic corticosteroids)
* Previous and / or current treatment with insulin (short term treatment due to intercurrent illness, including gestational diabetes, is allowed at the discretion of the investigator)
* Treatment with glucagon-like peptide-1 (GLP-1) receptor agonists, sulpfonylurea, glinides, dipeptidyl peptidase 4 (DPP-4) inhibitors or sodium-glucose co-transporter 2 (SGLT2) inhibitors within 90 days prior to the screening visit
* Impaired liver function, defined as alanine aminotransferase (ALAT) above or equal to 2.5 times upper normal range (UNR)
* Impaired renal function defined as serum-creatinine above or equal to 133 micromol/L (above or equal to 1.5 mg/dL) for males and above or equal to 125 micromol/L (above or equal to 1.4 mg/dL) for females, or as defined according to local contraindications for metformin
* Screening calcitonin above or equal to 50 ng/L
* Proliferative retinopathy or maculopathy (macular oedema) requiring acute treatment, according to investigator's clinical judgment
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2)
* History of pancreatitis (acute or chronic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2015-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (72):
- United States (37):
  - Novo Nordisk Investigational Site, Hamilton, Alabama
  - Novo Nordisk Investigational Site, Chandler, Arizona
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Hallandale, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Conyers, Georgia
  - Novo Nordisk Investigational Site, Blackfoot, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Crestview Hills, Kentucky
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Katy, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Austria (4):
  - Novo Nordisk Investigational Site, Linz
  - Novo Nordisk Investigational Site, Mödling
  - Novo Nordisk Investigational Site, St. Stefan
  - Novo Nordisk Investigational Site, Vienna
- Bulgaria (5):
  - Novo Nordisk Investigational Site, Kozloduy
  - Novo Nordisk Investigational Site, Lukovit
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Canada (8):
  - Novo Nordisk Investigational Site, Burnaby, British Columbia
  - Novo Nordisk Investigational Site, Coquitlam, British Columbia
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Moncton, New Brunswick
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Liverpool, Nova Scotia
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Waterloo, Ontario
- Czechia (4):
  - Novo Nordisk Investigational Site, Olomouc, Lazce
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Trutnov
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Szombathely
  - Novo Nordisk Investigational Site, Zalaegerszeg
- Russia (4):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Cheboksary
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Samara
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Slovakia (5):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Dunajská Streda
  - Novo Nordisk Investigational Site, Sabinov
  - Novo Nordisk Investigational Site, Vranov nad Topľou
  - Novo Nordisk Investigational Site, Žilina

REFERENCES:
- [Result] Safety and Efficacy of Insulin Degludec/Liraglutide(IDegLira) Titrated Once Weekly (1 Wk) vs. Twice Weekly (2 Wk) in Patients (pts) with T2D Uncontrolled on Oral Antidiabetic Drugs: DUAL VI Study; Stewart B. Harris et al. American Diabetes Association - 76th Annual Scientific Sessions; 10 June 2016
- [Result] Harris SB, Kocsis G, Prager R, Ridge T, Chandarana K, Halladin N, Jabbour S. Safety and efficacy of IDegLira titrated once weekly versus twice weekly in patients with type 2 diabetes uncontrolled on oral antidiabetic drugs: DUAL VI randomized clinical trial. Diabetes Obes Metab. 2017 Jun;19(6):858-865. doi: 10.1111/dom.12892. Epub 2017 Mar 3. PMID 28124817
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 80 sites in 9 countries as follows:Austria: 6 sites; Bulgaria: 5 sites; Canada: 7 sites, Czech Republic:5 sites; Hungary: 4 sites, Russian Federation: 6 sites; Serbia: 4sites, Slovakia: 7 sites; United States: 36 sites.
Pre-assignment Details: Stable daily treatment with metformin (≥1500 mg or max tolerated dose) ± pioglitazone (≥30 mg) for at least 90 days prior to screening
Groups:
- IDegLira (1WT): Subjects inadequately controlled on metformin either alone or in combination with pioglitazone were randomized in a 1:1 manner to receive IDegLira once daily. The subjects were stratified by their OAD treatment prior to entering the trial. The starting dose of IDegLira was 10 dose steps (10 units IDeg/0.36mg liraglutide), and the maximum dose was 50 dose steps (50units/1.8mg liraglutide) The daily dose for metformin was ≥ 1500mg or max tolerated dose and ≥ 30mg for pioglitazone. In the IDegLira once weekly titration group (1WT), the dose of IDegLira was adjusted based on the mean of 2 fasting SMPG values measured pre-breakfast in the morning of two consecutive days corresponding to one obtained on the day before titration and one obtained on titration day.
- IDegLira: Subjects inadequately controlled on metformin either alone or in combination with pioglitazone were randomized in a 1:1 manner to receive IDegLira once daily. The subjects were stratified by their OAD treatment prior to entering the trial. The starting dose of IDegLira was 10 dose steps (10 units IDeg/0.36mg liraglutide), and the maximum dose was 50 dose steps (50units/1.8mg liraglutide) The daily dose for metformin was ≥ 1500mg or max tolerated dose and ≥ 30mg for pioglitazone. In the IDegLira twice weekly titration group (1WT), the dose of IDegLira was adjusted based on the mean of 3 fasting SMPG values measured pre-breakfast in the morning of three consecutive days corresponding to one obtained on each of two days before titration and one obtained on titration day.
Period: Overall Study
Arm/Group | IDegLira (1WT) | IDegLira
Started | 210 | 210
Completed | 191 | 204
Not Completed | 19 | 6
Not completed — Unclassified | 3 | 2
Not completed — Withdrawal criteria | 2 | 0
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 6 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): Included all randomised subjects. The subjects in IDegLira (IWT) and IDegLira are 210 in each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegLira (1WT) | IDegLira | Total
Number analyzed (Participants) | 210 | 210 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10.3) | 57.0 (9.6) | 56.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 98 | 197
  Male | 111 | 112 | 223
HbA1c [Mean (Standard Deviation); unit: percentage] | 8.2 (0.9) | 8.1 (0.9) | 8.1 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c
Description: Change in glycosylated haemoglobin A1c (HbA1c) (%) from baseline after 32 weeks of treatment.
Time Frame: Week 0, week 32
Population: Full analysis set (FAS) included all randomised subjects. 20 subjects in the IDegLira (1WT) and 10 subjects in the IDegLira arm did not contribute to the analysis for this endpoint.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | IDegLira (1WT) | IDegLira
Number analyzed (Participants) | 189 | 200
percentage | -2.01 (1.09) | -2.02 (0.98)
Statistical Analysis 1: Comparison: IDegLira (1WT) vs IDegLira; The null hypothesis was tested against the alternative hypothesis of non-inferiority as given by H0: D ≥0.30% against HA: D <0.30%; Test type: Non-Inferiority or Equivalence — The null hypothesis was tested against the alternative hypothesis of non-inferiority as given by H0: D ≥0.30% against HA: D <0.30%; p = 0.012, Mixed Models Analysis; Treatment Contrast = 0.12, 95% CI 2-sided [-0.04 to 0.28]

2. Secondary Outcome: HbA1c Below 7.0%
Description: Responders to HbA1c below 7% after 32 weeks of treatment.
Time Frame: Week 0, week 32
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IDegLira (1WT) | IDegLira
Number analyzed (Participants) | 189 | 200
participants
  yes | 170 | 179
  No | 19 | 21

3. Secondary Outcome: HbA1c Below or Equal to 6.5%
Description: Responders to HbA1c below or equal to 6.5% after 32 weeks of treatment.
Time Frame: Week 0, week 32
Population: as for outcome 1
Measure: Number; unit: particpants
Arm/Group | IDegLira (1WT) | IDegLira
Number analyzed (Participants) | 189 | 200
particpants
  yes | 158 | 170
  No | 31 | 30

4. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: An episode that is severe according to the ADA classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 0-32
Population: Safety Analysis Set (SAS): Included all subjects receiving at least one dose of trial product. Subjects contributed to the evaluation "as treated". One subject in the IDegLira (1WT) arm did not contribute to the analysis for this endpoint.
Measure: Number; unit: Number of episodes
Arm/Group | IDegLira (1WT) | IDegLira
Number analyzed (Participants) | 209 | 210
Number of episodes | 20 | 97

ADVERSE EVENTS:
Time Frame: Defined as an event that has onset date on or after the first day of exposure to randomised treatment and no later than seven days after the last day of randomised treatment. (Visit 1- Visit 36)
Description: Safety Analysis Set (SAS): Included all subjects receiving at least one dose of trial product. Subjects contributed to the evaluation "as treated".
Groups:
- IDegLira (1WT): Subjects received IDegLira once weekly in combination with metformin alone or in combination with pioglitazone in a 1:1 manner at visit 2 and were stratified by their OAD treatment prior to entering the trial. The starting dose of IDegLira was 10 dose steps (10 units IDeg/0.36 mg liraglutide), and the maximum dose was 50 dose steps (50 units IDeg/1.8 mg liraglutide).The daily dose for metformin (≥1500 mg or max tolerated dose) and pioglitazone (≥30 mg) The dose of IDegLira was to be adjusted once weekly based on the mean of 2 fasting SMPG values measured pre-breakfast in the morning of two consecutive days corresponding to one obtained on the day before titration and one obtained on the titration day. The first dose of trial product was to be administered either on the day of randomisation (visit 2) or the day after.
Arm/Group | IDegLira (1WT) | IDegLira
Serious Adverse Events (participants affected / at risk) | 7/209 | 14/210
Other Adverse Events (participants affected / at risk) | 24/209 | 19/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (1WT) (N=209) | IDegLira (N=210)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (1WT) (N=209) | IDegLira (N=210)
Nasopharyngitis (Infections and infestations) | 13 (16) | 9 (13)
Nausea (Gastrointestinal disorders) | 11 (16) | 11 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator (s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for upto 60 days to protect intellectual property.